CLINICAL TRIAL: NCT05323617
Title: Two Arm Bridging Study to Evaluate the Efficacy of Romiplostim in the Treatment of Adult Severe Aplastic Anemia Participants Who Are Either Previously Untreated With IST or Refractory to IST
Brief Title: Efficacy of Romiplostim in Treatment of SAA in Adults Previously Untreated With or Refractory to Immunosuppressive Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Operational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210112
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Severe Aplastic Anemia; SAA; Very Severe Aplastic Anemia; vSAA; Romiplostim
MeSH Terms: conditions — Anemia, Aplastic | interventions — romiplostim; Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Previously Untreated IST (Experimental): Participants with SAA/vSAA that are previously untreated with IST.
  Interventions: Drug: Romiplostim; Drug: Antithymocyte Globulin; Drug: Cyclosporine A
- Arm 2: Refractory IST (Experimental): Participants with SAA/vSAA that are refractory to IST.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Administered as a subcutaneous injection.
  Other Names: Nplate®
Drug: Antithymocyte Globulin — Horse or rabbit antithymocyte globulin administered as an intravenous infusion.
  Arms: Arm 1: Previously Untreated IST
Drug: Cyclosporine A — Administered orally.
  Arms: Arm 1: Previously Untreated IST

SUMMARY:
Romiplostim has been used in clinical trials for the treatment of severe and very severe aplastic anemia (SAA/vSAA) in Asian participants who are either previously untreated with immunosuppressive therapy (IST) or refractory to IST. This study will evaluate the efficacy of romiplostim in the treatment of participants with SAA/vSAA.

The primary objectives of this study are to:

Arm 1: Evaluate the efficacy of romiplostim and IST in adult SAA/vSAA participants who are previously untreated with IST (1L)

Arm 2: Evaluate the efficacy of romiplostim treatment in adult SAA/vSAA participants who are refractory to IST (2L+)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of enrollment
* Diagnosis of SAA/vSAA confirmed by blood, bone marrow, and cytogenetic studies
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1 at screening
* Arm 1 only: participant requires initial treatment for SAA/vSAA, no matched related donor is available for allogenic hematopoietic cell transplantation (HCT) and will begin IST with antithymocyte globulin and CsA
* Arm 2 only: refractory to at least one course of immunosuppressive therapy including horse or rabbit ATG; or ineligible for ATG treatment and refractory to CsA

Exclusion Criteria:

* Diagnosed as having congenital aplastic anemia (AA) (Fanconi anemia, congenital dyskeratosis, etc)
* History of other malignancy within the past 5 years, with exceptions.
* Aplastic anemia with hemolytic paroxysmal nocturnal hemoglobinuria (PNH) (hemolytic predominant is defined as lactate dehydrogenase (LDH) > 1.5 x the upper limit of site normal
* Arm 1 only: Previously treated with ATG, CsA, or Alemtuzumab
* Previously treated with PEGylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), recombinant human thrombopoietin protein (TPO), romiplostim and other TPO-receptor agonist (eltrombopag, etc)
* Patients who are eligible for allogenic HCT and have an available matched related donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Arms 1 and 2: proportion of participants achieving any hematologic response at week 14 | Week 14
  Proportion of participants achieving any hematologic response at week 14 based on response criteria:
  * Platelet response
  * Erythroid response
  * Red blood cell count
  * Hemoglobin concentration
  * Neutrophil response

SECONDARY OUTCOMES:
Arm 1: number of participants who achieve a complete response (CR) or partial response (PR) at week 14 | Week 14
Arms 1 and 2: number of participants who have a decrease in frequency of platelet and/or red blood cell (RBC) transfusions, or become platelet and/or RBC transfusion independent at week 14 | Week 14
Arms 1 and 2: number of participants with serious adverse events | 24 Weeks
Arms 1 and 2: number of participants with clinically significant changes in laboratory values | 24 Weeks
Arms 1 and 2: change from baseline in Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto (GIMEMA) bleeding scale at week 14 | Baseline and Week 14
  The Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto is as follows:
  0: No bleeding
  1. Petecjoae or mucosal or retinal bleeding that did not require red-cell transfusion
  2. Melena, hematemesis, hematuria, or hemoptysis
  3. Any bleeding that required red-cell transfusion
  4. Retinal bleeding accompanied by visual impairment
  5. Nonfatal cerebral bleeding
  6. Fatal cerebral bleeding
  7. Fatal noncerebral bleeding
Arms 1 and 2: serum romiplostim trough concentrations | Prior to romiplostim administration on Weeks 1, 2, 4, 5, 9, 13, and 24
Arms 1 and 2: maximum serum concentration (Cmax) of romiplostim | Weeks 1, 2, 4, 5, 9, 13, and 24
Arms 1 and 2: area under the curve (AUC) of romiplostim | Weeks 1, 2, 4, 5, 9, 13, and 24
Arms 1 and 2: time to reach maximum concentration (tmax) of romiplostim | Weeks 1, 2, 4, 5, 9, 13, and 24
Arms 1 and 2: half-life (t1/2) of romiplostim | Weeks 1, 2, 4, 5, 9, 13, and 24
Arms 1 and 2: number of participant with anti-romiplostim antibodies | Prior to romiplostim administration on Weeks 1 and 13
Arms 1 and 2: number of participants with antibodies to thrombopoietin | Prior to romiplostim administration on Weeks 1 and 13

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com